CLINICAL TRIAL: NCT02537821
Title: HLA Sensitization in Severely Burned Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: PKSF-01-2014
Record Dates: First submitted 2015-07-01; First posted 2015-09-02 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Severely Burned Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Primary goal of this study is the analysis of HLA (Human leucocyte antigen) formation in severly burned patients. Potential HLA triggers in the treatment of severely burned patients are blood products, assist devices or temporary allogeneic skin. Besides that, inflammatory markers, such as WBC (white blood cell count), CRP (C-reactive protein), PCT (Procalcitonin) and two novel biomarkers (PSP (pancreatic stone protein), ST2) are to be investigated in severely burned patients.

ELIGIBILITY:
Inclusion Criteria:

* severely burned patients in need for hospitalization

Exclusion Criteria:

* hematologic diseases
* Cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severely burned patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
HLA antibody formation (HLA Sensitization) (Unit: PRA in %) | Change from Baseline (admission) in HLA antibody count at 2 weeks, 4 weeks, 3 months and 6 months
  The degree of sensitization is reported as the percentage of CDC (Complement dependent Cytotoxicity) Panel Reactive Antibody (PRA). Unit is %.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Plock, M.D., Principal Investigator — Raemistrasse 100, 8091
Locations (1):
- University Hospital Zurich, Zurich, Switzerland